CLINICAL TRIAL: NCT05446168
Title: Brain Small Chain Fatty Acid Metabolism in Parkinson Disease: Tributyrin Supplementation
Acronym: BUTTER
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: Nicolaas Bohnen, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Nicolaas Bohnen, MD, PhD, Professor of Radiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00211320
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: short chain fatty acid; butyrate; tributyrin; functional neuroimaging
MeSH Terms: conditions — Parkinson Disease | interventions — tributyrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parkinson's Disease Tributyrin Intervention (Experimental): Participants will take 500mg TID tributyrin supplement for 30 days +/- 7 days.
  Interventions: Drug: tributyrin
- Healthy Control Tributyrin Intervention (Experimental): Participants will take 500mg TID tributyrin supplement for 30 days +/- 7 days.
  Interventions: Drug: tributyrin

INTERVENTIONS:
Drug: tributyrin — Post-biotic short chain fatty acid dietary supplement. Participants will take 500mg TID tributyrin supplement for 30 days +/- 7 days.

SUMMARY:
Small exploratory open-label pilot study to assess the short-chain fatty acid (SCFA) prodrug tributyrin as a potential therapy for persons with Parkinson disease

DETAILED DESCRIPTION:
The overarching goal of this small exploratory open-label pilot study is to explore metabolic (glucose metabolism, butyrate) and cognition (MoCa) before and after open-label treatment with the short-chain fatty acid (SCFA) prodrug tributyrin in a small pilot study in PD and normal control older adults. Positive findings in this small exploratory pilot trial may support target engagement study of SCFA supplementation in normal adults and PD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control volunteers over 45 years of age
* People with Parkinson Disease over 45 years of age

Exclusion Criteria:

* Subjects with contra-indications to MR imaging, including pacemakers or claustrophobia;
* Evidence of large vessel stroke or mass lesion on MRI
* Regular use of anti-cholinergic, benzodiazepines or neuroleptic drugs
* History of significant GI disease
* Significant metabolic or uncontrolled medical comorbidity
* Poorly controlled diabetes
* Pregnancy or breast feeding
* Dementia requiring informed assent
* Suicidal ideation

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas I Bohnen, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System Functional Neuroimaging, Cognitive and Mobility Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 participants were enrolled in the study. One Parkinson's disease subject withdrew prior to beginning study procedures and thus is not counted as started.
Period: Overall Study
Arm/Group | Parkinson's Disease Tributyrin Intervention | Healthy Control Tributyrin Intervention
Started | 14 | 3
Completed | 14 | 2
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease Tributyrin Intervention | Healthy Control Tributyrin Intervention | Total
Number analyzed (Participants) | 14 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 9 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (5.7) | 67.3 (10.6) | 66.5 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 9 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 3 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 3 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 3 | 16
Education [Mean (Standard Deviation); unit: years] | 17.9 (2.8) | 19.3 (3.5) | 18.1 (2.9)
Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III [Mean (Standard Deviation); unit: units on a scale] — The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 3 is a clinician-administered motor exam consisting of 18 items to evaluate the motor symptom severity in Parkinson's disease. Total scores range from 0 to 132, with higher scores indicating higher severity of motor symptoms. MDS-UPDRS Part 3 scores of 32 and below are typically considered mild, 33-58 is moderate, and 59 and above considered severe.
  units on a scale | 46.9 (12.7) | 28.0 (20.5) | 43.6 (15.5)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is used for detection of mild cognitive impairment. It assesses short-term memory, visuospatial abilities, executive functioning, attention, language, and orientation. Scores range from 0 to 30, with low scores indicating more cognitive impairment. Scores of 26 and above indicate normal cognitive performance, 18-25 indicate mild impairment, 10-17 indicate moderate impairment, and 0-9 indicate severe impairment.
  units on a scale | 26.8 (2.9) | 27.7 (1.2) | 26.9 (2.7)
Parkinson's Disease Cognitive Rating Scale (PDCRS) [Mean (Standard Deviation); unit: units on a scale] — The Parkinson's Disease Cognitive Rating Scale (PDCRS) evaluates cognition in Parkinson's disease. Scores range from 0-134 with lower scores indicating increased cognitive impairment.
  units on a scale | 92.0 (12.3) | 96.3 (3.8) | 92.8 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Whole Brain Butyrate PET Radiotracer Binding
Description: Whole-brain butyrate distribution volume ratios (DVRs) were computed relative to a cerebral white matter reference region pre and post approximately 30 days of open-label treatment with tributyrin. Lower radiotracer binding is interpreted to reflect higher levels of (non-tracer) butyrate in the brain, whereas higher radiotracer binding reflects higher butyrate receptor binding site availability, indicating lower levels of non-tracer butyrate in the brain.
Time Frame: Pre and Post approximately 30 days of intervention
Population: Brain imaging was not strictly required for participation in the remaining components of the study. Not all participants underwent PET imaging. Healthy control sample size (n=2) was not sufficient to perform statistical analysis for that group.
Measure: Mean (Standard Deviation); unit: Parametric DVR
Arm/Group | Parkinson's Disease Tributyrin Intervention | Healthy Control Tributyrin Intervention
Number analyzed (Participants) | 8 | 2
Parametric DVR
  Pre-intervention | 1.81 (0.10) | 1.79 (0.02)
  Post-intervention | 1.73 (0.10) | 1.74 (0.01)
Statistical Analysis 1: Comparison: Parkinson's Disease Tributyrin Intervention; Test type: Other — A comparison is not being made between two different treatment groups. Exploratory analysis; p = 0.005, t-test, 2 sided — A priori threshold for statistical significance is p < 0.05; t = -4.05, df = 7; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.12 to -0.03], Standard Deviation 0.05

2. Primary Outcome: Glucose Metabolism
Description: Continuous glucose meter 7-10-day average glucose readings before/after open-label treatment with the SCFA prodrug tributyrin in patients with PD and normal controls. Healthy fasting blood glucose ranges from 70 to 99 milligrams per deciliter (mg/dL), with a healthy maximum of 180 mg/dL withing 2 hours of eating meals.
Time Frame: Pre and Post approximately 30 days of intervention
Population: 2 Parkinson's disease participants did not complete continuous glucose monitoring due to scheduling conflicts, thus only 14/16 participants were included in this analysis. Healthy control sample size (n=2) was not sufficient to perform statistical analysis for that group.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Parkinson's Disease Tributyrin Intervention | Healthy Control Tributyrin Intervention
Number analyzed (Participants) | 12 | 2
milligrams per deciliter (mg/dL)
  Pre-Intervention | 135.00 (49.39) | 104.50 (3.54)
  Post-Intervention | 139.33 (53.31) | 125.00 (4.24)
Statistical Analysis 1: Comparison: Parkinson's Disease Tributyrin Intervention; Test type: Other — A comparison is not being made between two different treatment groups. Exploratory analysis; p = 0.27, t-test, 2 sided — A priori threshold for statistical significance is p < 0.05; t = 1.17, df = 11; Mean Difference (Net) = 4.33, 95% CI 2-sided [-3.81 to 12.47], Standard Deviation 12.81

ADVERSE EVENTS:
Time Frame: For all subjects, data was collected during the 30 +/- 7 days of tributyrin intervention.
Arm/Group | Parkinson's Disease Tributyrin Intervention | Healthy Control Tributyrin Intervention
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/3
Other Adverse Events (participants affected / at risk) | 13/14 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson's Disease Tributyrin Intervention (N=14) | Healthy Control Tributyrin Intervention (N=3)
GI Discomfort (Gastrointestinal disorders) | 7 (8) | 0 (0) — Related, mild, expected AE
Behavioral Disturbance (Psychiatric disorders) | 0 (0) | 1 (1) — Unrelated, mild, unexpected AE
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Unrelated, mild, unexpected AE
Sleep Disruption (Nervous system disorders) | 3 (3) | 0 (0) — Unrelated, mild, unexpected AE
Shakiness/Dyskinesia (Nervous system disorders) | 2 (2) | 0 (0) — Unrelated, mild, unexpected AE
Toe Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated, mild, unexpected AE
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0) — Unrelated, mild, unexpected AE
Respiratory Infection (Infections and infestations) | 4 (4) | 0 (0) — Unrelated, mild, unexpected AE
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) — Unrelated, mild, unexpected AE
Gait Disturbances (Nervous system disorders) | 1 (1) | 0 (0) — Unrelated, mild, unexpected AE
Leg Swelling (Vascular disorders) | 1 (1) | 0 (0) — Unrelated, mild, unexpected AE
High Blood Glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Unrelated, mild, unexpected AE
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Unrelated, mild, unexpected AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT05446168/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT05446168/ICF_000.pdf